CLINICAL TRIAL: NCT06766487
Title: Chang Gung Memorial Hospital At Linkou
Brief Title: Effectiveness of Tongue Resistance Exercises on Tongue and Swallowing Function in Frail Older Adults with MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Medical Foundation (Other)
Collaborators: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Kao, Shu-Hua, Chang Gung Medical Foundation, Chang Gung Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202001044; CMRPG5L0032 (Other Grant/Funding Number: Chang Gung Memorial Hospital at Linkou)
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2023-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Tongue Resistance Exercises; Frail; Swallowing Function
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The experimental group performed tongue resistance exercises, while the control group practiced cheek bulging exercises.
  This study adopts a longitudinal research design with randomization. Participants were randomly assigned to two groups using an online computer-based randomization tool.
Who Masked: Participant, Care Provider
Masking Description: This study employed a prospective, double-blind, randomized controlled trial design to investigate the effects of TREs in frail older adults with MCI. Potential participants from nursing homes and community-based daytime long-term care centers underwent eligibility screening. To ensure blinding, a research assistant not directly involved in the study conducted random sequence generation for group allocation using an online computer-based randomization program. Block randomization (1:1 ratio) was implemented to maintain equal group sizes. The research assistant then sealed the group allocation data in opaque envelopes, which were stored securely in a locked cabinet. Both participants and researchers were blinded to group assignment. Participants remained unaware of their assigned intervention (TREs or cheek-bulging exercises), and researchers were also blinded to participant group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tongue Resistance Exercises (Experimental): TRTP involved movements of the tongue's anterior, middle, posterior, and lateral parts, targeting the intrinsic and extrinsic tongue muscles and the soft palate.
  Interventions: Behavioral: Tongue resistance exercises
- cheek bulging exercises (Placebo Comparator): Cheek bulging exercises involved closing the lips, bulging the right cheek, relaxing and returning to the initial position, bulging the left cheek, relaxing and returning to the initial position, and finally bulging both cheeks simultaneously.
  Interventions: Behavioral: cheek bulging exercises

INTERVENTIONS:
Behavioral: Tongue resistance exercises — The TRE program consisted of the following exercises:
  Exercise 1: Tongue Protrusion and Retraction Against Resistance, Exercise 2: Anterior Tongue Protrusion and Retraction Against Resistance, Exercise 3: Middle Tongue Protrusion and Retraction Against Resistance, Exercise 4: Middle Tongue Elevation with Pharyngeal Sound Production, Exercise 5: Tongue Elevation and Posterior Sweeping, and Exercise 6: Saliva Swallowing with Lip Closure.
  Arms: Tongue Resistance Exercises
Behavioral: cheek bulging exercises — Cheek bulging exercises involved a series of movements: Lip Closure: Participants began by closing their lips. Unilateral Cheek Bulging: They then bulged their right cheek, followed by relaxation and return to the initial position. This was repeated on the left side. Bilateral Cheek Bulging: Finally, participants bulged both cheeks simultaneously.
  Arms: cheek bulging exercises

SUMMARY:
The purpose of this study is to explore the effects of tongue resistance exercises on tongue muscle strength and swallowing function in frail older adults with mild cognitive impairment living in the community.

This study adopts a longitudinal research design with randomization. Participants were randomly assigned to two groups using an online computer-based randomization tool. The experimental group performed tongue resistance exercises, while the control group practiced cheek bulging exercises.

DETAILED DESCRIPTION:
Recruitment took place in nursing homes, day care centers, and community care centers across Taiwan. Participants were older adults aged 65 years or older with mild cognitive impairment and frailty, enrolled between August 1, 2021, and July 31, 2022.

Participants were randomly divided into two groups by computer, 23 peoples per group, The experimental group performed tongue resistance exercises, while the control group practiced cheek bulging exercises. The exercise intervention is 12 weeks of exercise begins, with each session 30 minutes.

The evaluation items include basic information, outcomes collected through a Iowa Oral Performance Instrument (IOPI) was used to measure tongue strength, tongue endurance, tongue endurance time, saliva swallowing pressure, effortful saliva swallowing pressure, and Aspiration assessment. The measurement times are as follows: T0 (Baseline), T1 (Week 4, Mid-Intervention), T2 (Immediate Post-Test after the 12-Week Intervention), and T3 (Follow-Up after the 12-Week Intervention).

Before conducting the study, all participants received a complete explanation of the purpose, risks, and procedures of the investigation, and provided written informed consent. Procedures were in accordance with the ethical standards of the committee on human experimentation at the institution where the work was conducted, and this study was approved by the Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment in older adults aged ≥65 years
* Frailty assessment: at least 1 point

Exclusion Criteria:

* Having aspiration pneumonia
* Tracheotomy is retained

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Tongue strength (anterior tongue strength [ATS] and posterior tongue strength [PTS]) | Assessments were performed at baseline (T0), 4-week mid-intervention (T1), 12-week immediate post-intervention (T2), and 12-week follow-up (T3).
  Tongue strength was measured using IOPI (Model 3.1) device, which was set to record peak pressure and repeated strength to evaluate the maximum pressure exerted during each repetition . The bulb was placed on the palate inside the upper front teeth and at the junction of the hard palate and soft palate to measure ATS and PTS. Maximum isometric pressure (MIP) was defined as the pressure generated when the participant pushed the tongue forcefully against the palate and maintained it for 3 seconds for both the anterior and posterior tongue. Each exercise was performed thrice, with 1-minute intervals between trials. The highest value from the three trials was recorded. MIP is reported in terms of kilopascals. The average pressure values for the anterior and posterior parts of the tongue were 55.95 ± 14.13 kPa and 53.23 ± 12.24 kPa, respectively.
Tongue Endurance (anterior tongue endurance [ATE] and posterior tongue endurance [PTE]) | Assessments were performed at baseline (T0), 4-week mid-intervention (T1), 12-week immediate post-intervention (T2), and 12-week follow-up (T3).
  Tongue endurance was measured using IOPI (Model 3.1) device using the target mode with the target value set at 50% of the individual's MIP. The bulb was placed on either the anterior tongue or the posterior tongue to measure ATE and PTE. The participant pushed the tongue against the palate for 3 seconds. If the pressure exceeded the target value, the instrument displayed a green light indicating the goal had been achieved. Tongue endurance was assessed only once. For the assessment of tongue endurance, interrater reliability was .97, and interrater reliability was .95. Tongue weakness, defined as a tongue pressure of <30 kPa, is associated with a risk of malnutrition.At the indicated cutoff values, the assessment sensitivity was 92% (95% CI: 75% to 98%), specificity was 96% (95% CI: 87% to 99%), positive predictive value was 92% (95% CI: 75% to 98%), negative predictive value was 96% (95% CI: 87% to 99%), and accuracy was 94.7% (95% CI: 87% to 98%).
Swallowing pressure (saliva swallowing pressure [SSP] and effortful swallow pressure [ESP]). | Assessments were performed at baseline (T0), 4-week mid-intervention (T1), 12-week immediate post-intervention (T2), and 12-week follow-up (T3).
  Saliva swallowing pressure (SSP) was measured using IOPI (Model 3.1). The IOPI device was set to record peak pressure and repeated strength to evaluate the maximum pressure exerted during each repetition. The bulb was placed on the palate inside the upper front teeth. The participant gently closed the mouth and then swallowed saliva normally (without pressing the bulb with the tongue). An SSP of <10.3 kPa among older adults is associated with an increased risk of aspiration pneumonia.Effortful Swallowing Pressure (ESP) was measured using IOPI (Model 3.1). The IOPI device was set to record peak pressure and repeated strength to evaluate the maximum pressure exerted during each repetition. The bulb was placed on the palate inside the upper front teeth. The participant gently closed the mouth performed an effortful saliva swallow (eg, an egg), but did not press the bulb with the tongue.
Aspiration assessment | Assessments were performed at baseline (T0), 4-week mid-intervention (T1), 12-week immediate post-intervention (T2), and 12-week follow-up (T3).
  The references were developed using a structured evaluation form. Information for each option was obtained by interviewing the case or caregiver or by reviewing the institution's records. The evaluation included determining whether there had been a physician-diagnosed case of pneumonia, a fever ≥ 38℃, or respiratory symptoms such as coughing or difficulty breathing, as well as recording the dates of occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Kao S Hua, Master, Study Chair — Chang Gung Medical Foundation Chang Gung Memorial Hospital at Linkou, Taoyuan, Taiwan
Locations (1):
- Chang Gung Memorial Hospital at Linkou, Taoyuan District, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leira J, Maseda A, Lorenzo-Lopez L, Cibeira N, Lopez-Lopez R, Lodeiro L, Millan-Calenti JC. Dysphagia and its association with other health-related risk factors in institutionalized older people: A systematic review. Arch Gerontol Geriatr. 2023 Jul;110:104991. doi: 10.1016/j.archger.2023.104991. Epub 2023 Mar 7. PMID 36906939
- [Background] Namiki C, Hara K, Tohara H, Kobayashi K, Chantaramanee A, Nakagawa K, Saitou T, Yamaguchi K, Yoshimi K, Nakane A, Minakuchi S. Tongue-pressure resistance training improves tongue and suprahyoid muscle functions simultaneously. Clin Interv Aging. 2019 Mar 22;14:601-608. doi: 10.2147/CIA.S194808. eCollection 2019. PMID 30962680
- [Background] Kim HD, Choi JB, Yoo SJ, Chang MY, Lee SW, Park JS. Tongue-to-palate resistance training improves tongue strength and oropharyngeal swallowing function in subacute stroke survivors with dysphagia. J Oral Rehabil. 2017 Jan;44(1):59-64. doi: 10.1111/joor.12461. PMID 27883209
- [Derived] Kao SH, Chen R, Su PY, Banda KJ, Sung CM, Wang CH, Chiang KJ, Fajarini M, Chou KR. A tongue resistance training program improves strength, endurance, and swallowing in frail older adults with mild cognitive impairment: a double-blind randomized controlled trial. Geroscience. 2025 May 29. doi: 10.1007/s11357-025-01715-5. Online ahead of print. PMID 40439971